CLINICAL TRIAL: NCT07233148
Title: Healing ALS Registry Observational Study (HAROS)
Acronym: HAROS
Status: Recruiting | Type: Observational
Sponsor: Healing Advocates Registry and Ministry (Other)
Responsible Party: Principal Investigator, William Lee Cowden, Principal Investigator, Healing Advocates Registry and Ministry
Other Study IDs: 25-12-299-2201
Record Dates: First submitted 2025-08-07; First posted 2025-11-18 (Actual); Last update posted 2026-01-28 (Actual); Status verified 2026-01

CONDITIONS: Amyotrophic Lateral Sclerosis (ALS); Motor Neuron Disease (MND); Primary Lateral Sclerosis (PLS)
Keywords: ALS; PLS; MND; Amyotrophic Lateral Sclerosis; Primary Lateral Sclerosis; Motor Neuron Disease; Motor Neurone Disease
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis; Motor Neuron Disease | interventions — Minerals; Meditation; Psychotherapy; Diet; Exercise; Physical Therapy Modalities; Occupational Therapy; Speech Therapy; Steam Bath; Massage; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- ALS/MND less than 3 years since diagnosis: Those diagnosed with ALS, Amyotrophic Lateral Sclerosis or MND, Motor Neuron Disease (other countries) and time since diagnosis is less 3 years, or 36 months, as of the date they join the study.
  Interventions: Other: Education about treatment options; Dietary Supplement: Dietary Supplements: Vitamins, Minerals, Herbs, etc.; Behavioral: Meditation, Prayer, Talk Therapy, Affirmations, Journaling, etc.; Other: Diet, various diets will be observed; Other: Exercise, physical therapy, occupational therapy, speech therapy, sauna, EMS, massage and other therapies; Drug: ALS medications and other medications; Other: Physical and emotional support
- PLS less than 3 years since diagnosis: Those diagnosed with PLS, Primary Lateral Sclerosis, and time since diagnosis is less 3 years, or 36 months, as of the date they join the study.
  Interventions: Other: Education about treatment options; Dietary Supplement: Dietary Supplements: Vitamins, Minerals, Herbs, etc.; Behavioral: Meditation, Prayer, Talk Therapy, Affirmations, Journaling, etc.; Other: Diet, various diets will be observed; Other: Exercise, physical therapy, occupational therapy, speech therapy, sauna, EMS, massage and other therapies; Drug: ALS medications and other medications; Other: Physical and emotional support
- ALS/MND 3 years or greater since diagnosis: Those diagnosed with ALS, Amyotrophic Lateral Sclerosis or MND, Motor Neuron Disease (other countries) and time since diagnosis is 3 years or greater as of the date they join the study.
  Interventions: Other: Education about treatment options; Dietary Supplement: Dietary Supplements: Vitamins, Minerals, Herbs, etc.; Behavioral: Meditation, Prayer, Talk Therapy, Affirmations, Journaling, etc.
- PLS 3 years or greater since diagnosis.: Those diagnosed with PLS, Primary Lateral Sclerosis and time since diagnosis is 3 years or greater as of the date they join the study.
  Interventions: Other: Education about treatment options; Dietary Supplement: Dietary Supplements: Vitamins, Minerals, Herbs, etc.; Behavioral: Meditation, Prayer, Talk Therapy, Affirmations, Journaling, etc.

INTERVENTIONS:
Other: Education about treatment options — Education about treatment options and integrative therapies is optional. It is available online and is free for all study participants.
Dietary Supplement: Dietary Supplements: Vitamins, Minerals, Herbs, etc. — The investigators are observing type and quantity of dietary supplements, vitamins, minerals and herbs that ALS/MND/PLS patients take regularly.
Behavioral: Meditation, Prayer, Talk Therapy, Affirmations, Journaling, etc. — Many of those diagnosed with ALS/MND/PLS regularly engage in meditation, prayer and other behavioral protocols. These will be observed and analyzed to see if, and to what degree they affect outcomes.
Other: Diet, various diets will be observed — May ALS/MND/PLS patients follow a specific diet such as ketogenic, vegetarian, gluten-free, dairy-free, and/or sugar-free. The investigators will analyze which diets are most efficacious.
  Groups: ALS/MND less than 3 years since diagnosis; PLS less than 3 years since diagnosis
Other: Exercise, physical therapy, occupational therapy, speech therapy, sauna, EMS, massage and other therapies — Exercise, physical therapy, occupational therapy, speech therapy, sauna, massage, EMS (electro-muscular stimulation), red light therapy and other physical modalities will be observed and analyzed for effect on outcomes.
  Groups: ALS/MND less than 3 years since diagnosis; PLS less than 3 years since diagnosis
Drug: ALS medications and other medications — Many ALS/MND/PLS patients find benefit from prescription and other drugs. These will be observed and analyzed for effect on quality of life and outcomes.
  Groups: ALS/MND less than 3 years since diagnosis; PLS less than 3 years since diagnosis
Other: Physical and emotional support — Study participants are asked to record the level of emotional and physical support they get from family members, caregivers, friends, medical professionals and members of their community. The investigators will analyze how the perceived level of emotional and physical support affect outcomes.
  Groups: ALS/MND less than 3 years since diagnosis; PLS less than 3 years since diagnosis

SUMMARY:
This is a prospective, observational, online study of people diagnosed with ALS, MND or PLS referred to as HAROS (Healing ALS Registry Observational Study). Participants will enter information into an online ALS registry once per month, including their ALSFRS-R data, certain other symptoms, dietary intake, supplements, medications and other therapies, both conventional and integrative. Participants will also enter the hours spent on optional self-study and free online education. The investigators will assess the effectiveness of various therapies and education by measuring physical outcomes.

DETAILED DESCRIPTION:
There is strong evidence that Amyotrophic Lateral Sclerosis (ALS), Motor Neuron Disease (MND) and Primary Lateral Sclerosis (PLS) are potentially reversible and NOT uniformly-fatal conditions, as reported in the literature. A 12-month 2024 retrospective, observational registry data analysis of 45 ALS patients showed that 85% did better than predicted in the peer-reviewed published literature. In fact, 20% did not lose functionality and 20% actually improved functional status over 12 months.

This prospective study seeks to enroll at least 1000 patients diagnosed with ALS, MND or PLS confirmed by their neurologist into this fully-remote, larger, observational study to see if the results of the 45-person ALS data analysis can be substantiated with a larger number of ALS, MND and PLS participants. Participants will be from the USA and other countries. In addition to that primary purpose, the investigators expect to:

* determine the efficacy of an integrative medicine approach to ALS (integrative medicine includes conventional medicine, functional medicine and other medical approaches such as acupuncture, frequency medicine and meditation)
* assess the effectiveness of self-study and integrative medicine education programs on ALS outcomes
* track data to analyze the most effective treatment protocols that ALS patients are currently engaged in and correlate with clinical outcomes
* explore and analyze possible causative factors and their treatments on outcomes using advanced data analysis

Study participants commit to updating their information monthly into the online registry for at least one year, preferably for up to 10 years. This takes approximately one hour per month. Participants choose their own treatment protocols based on their own research and input from their healthcare practitioners. Self-study and integrative medicine education is optional but encouraged. Participants in this study can join other research studies at the same time as HAROS, as long as they record in the registry all studies in which they are participating.

This study (HAROS) has the potential to improve the prognosis of patients with a diagnosis of ALS, MND or PLS when results are periodically shared about the effectiveness of various treatments and education.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with ALS, MND or PLS

Exclusion Criteria:

* Smokers

Ages: 18 Years to 110 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators are studying adult non-smokers who have a diagnosis of ALS, MND or PLS, irrespective of time since diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2026-01-26 (Actual); Primary Completion 2036-02-05 (Estimated); Study Completion 2036-03-31 (Estimated)

PRIMARY OUTCOMES:
ALSFRS-R ALS Functional Rating Scale - Revised | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  ALS Functional Ratings Scale is a set of 12 questions, with a maximum of 4 points per question and measures physical functionality. Outcomes are measured at a point in time and range from 0 for no functionality to 48 for full functionality in all areas measured. The higher the score the better the outcome.
ALSSQ ALS Supplementary Questionnaire | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  ALS Supplementary Questionnaire (ALSSQ) is a measure of physical functionality and symptoms that are not measured in the ALSFRS-R scale. Items measured in the ALSSQ are energy level, sleep quality and quantity, pain, fasciculations, muscle cramps, mucous, mental clarity, head drop and showing emotions inappropriately. There are 18 questions, 4 points each, for a maximum of 72 points. The higher this score, the better the outcome.
Mindset Score | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  Mindset is measured by questions about A) positivity, maximum 400 points, B) belief in ability to get well and mental blocks to healing, maximum 18 points, and C) a Modified PANAS (Positive and Negative Affect Schedule), maximum of 50 positive points and 50 negative points. The investigators will analyze how these measures of mindset correlate with ALS/MND/PLS outcomes.

SECONDARY OUTCOMES:
Weight | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  Body Weight is often an issue with ALS/MND/PLS patients. The investigators will observe any correlation between body weight and outcomes.
Change in blood inflammation markers Set 1 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician and recorded.
  Inflammation and neuroinflammation are often associated with ALS/MND/PLS. Higher inflammatory markers may be correlated with faster disease progression. The investigators will analyze how these measures correlate with ALS/MND/PLS outcomes.
  NfL plasma (Neurofilament Light chain - plasma) pg/mL NfL serum (Neurofilament Light chain - serum) pg/mL Interleukin-6 pg/ml TMAO (Trimethylamine-N-Oxide) pg/mL
Change in blood inflammation markers Set 2 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician and recorded.
  Inflammation and neuroinflammation are often associated with ALS/MND/PLS. Higher inflammatory markers may be correlated with faster disease progression. The investigators will analyze how these measures correlate with ALS/MND/PLS outcomes.
  hs-CRP (high sensitivity C-Reactive Protein) mg/dL GGT (gamma-glutamyl transferase) mg/dL
Change in blood oxidative stress markers Set 1 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Higher oxidative stress may be correlated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  1. Serum Ferritin measured in ng/ml
  2. oxLDL (oxidized LDL) measured in ng/ml
  3. Serum 8-OHdG (8-hydroxy-2-deoxyguanosine) measured in ng/ml
Change in blood oxidative stress markers Set 2 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Higher oxidative stress may be correlated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  a. Serum malondialdehyde measured in nmol/mL
Change in blood essential nutrient levels Set 1 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Levels of essential nutrients may be associated with faster or slower disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  1. RBC magnesium (mg/dL)
  2. Ceruloplasmin (mg/dL)
Change in blood essential nutrient levels Set 2 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Levels of essential nutrients may be associated with faster or slower disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  a. Vitamin D-25 Hydroxy (ng/mL)
Change in blood essential nutrient levels Set 3 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Levels of essential nutrients may be associated with faster or slower disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  1. Arachidonic Acid (µg/mL)
  2. Alpha-Linolenic Acid (µg/mL)
  3. Linoleic Acid (µg/mL)
  4. DGLA (Dihomo-gamma-linolenic acid) (μg/mL)
  5. EPA (Eicosapentaenoic acid) μg/mL
  6. DHA (Docosahexaenoic acid) μg/mL
Change in blood essential nutrient levels Set 4 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Levels of essential nutrients may be associated with faster or slower disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  1. Methylmalonic acid (μmol/L)
  2. Serum Homocysteine (μmol/L)
Change in blood essential nutrient levels Set 5 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Levels of essential nutrients may be associated with faster or slower disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  1. Vitamin A Retinol (μg/dL)
  2. Serum Copper (μg/dL)
  3. Serum Zinc (μg/dL)
Change in blood insulin resistance markers Set 1 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Insulin resistance may be correlated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  1. Insulin, fasting (mg/dL) (higher indicates higher level of insulin resistance)
  2. Blood Glucose, fasting (mg/dL) (higher indicates higher level of insulin resistance)
  3. Triglycerides (mg/dL) (higher indicates higher level of insulin resistance)
Change in blood insulin resistance markers Set 2 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Insulin resistance may be correlated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  a. HDL Cholesterol (mg/dL) (lower indicates higher level of insulin resistance)
Change in blood insulin resistance markers Set 3 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Insulin resistance may be correlated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  a. Fructosamine, fasting (µmol/L) (higher indicates higher level of insulin resistance)
Change in blood insulin resistance markers Set 4 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Insulin resistance may be correlated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  a. Hemoglobin A1C (percent) (higher indicates higher level of insulin resistance)
Change in blood infection markers Set 1 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Infection markers in the blood may be associated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes. A higher IgG indicates a higher level of infection.
  1. IgG to Epstein Barr Viral Capsid Antigen (U/mL))
  2. IgG to Epstein Barr Nuclear Antigen (U/mL)
Change in blood infection markers Set 2 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Infection markers in the blood may be associated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes. A higher titer indicates a higher level of infection.
  1. IgG to HHV-6 Viral Antigen (Human Herpes Virus type 6) (titer)
  2. IgG to Coxsackie B virus Antigen (titer)
  3. Poliovirus Type 1 Antibodies (titer)
  4. Poliovirus Type 3 Anitbodies (titer)
Change in blood infection markers Set 3 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Infection markers in the blood may be associated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate withALS/MND/PLS outcomes. The higher the marker, the higher the level of infection.
  1. WBC (White Blood Cells) (k/uL)
  2. Neutrophils (k/uL) cells per microliter in thousands
  3. Lymphocytes (k/uL) cells per microliter in thousands
  4. CD57 (k/uL) cells per microliter in thousands
Change in blood infection markers Set 4 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Infection markers in the blood may be associated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes. A higher C4A can indicate a higher level of infection, inflammation or autoimmune conditions.
  a. C4A (Complement 4A) (mg/dL)
Change in blood infection markers Set 5 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Infection markers in the blood may be associated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes. A higher LPS can indicate bacteria from the gut entering the bloodstream because of increased intestinal permeability.
  a. LPS Lipopolysaccharides by Endotoxin Activity Assay (EU - Endotoxin Units)
Change in urine toxin markers Set 1 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Increased levels of urine toxins may be associated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  1. Urine aflatoxin (ppb)
  2. Urine gliotoxin (ppb)
  3. Urine trichothecene (ppb)
Change in urine toxin markers Set 2 | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician. Increased levels of urine toxins may be associated with faster disease progression of ALS/MND/PLS. The investigators will analyze how a change in these measures correlate with ALS/MND/PLS outcomes.
  1. Urine mercury (µg/L)
  2. Urine lead (µg/L)
Change in NfL (Neurofilament Light chain) | Participants will be assessed at baseline and each 1 year anniversary from the baseline until participant withdraws from the study for any reason, including death from any cause, up to a maximum of 10 years from baseline.
  All lab tests are optional, and ordered through the patient's physician and recorded. NfL (lNeurofilament Light chain) can be used to assess neuronal damage with ALS/MND/PLS. A higher level of NfL often indicates a higher level of neuronal damage. The investigators will analyze how changes in NfL correlate with ALS/MND/PLS outcomes.
  1. NfL plasma (Neurofilament Light chain - plasma) pg/mL
  2. NfL serum (Neurofilament Light chain - serum) pg/mL

CONTACTS AND LOCATIONS:
Overall Officials: William L Cowden, MD, Principal Investigator — Chair of Scientific Board of Academy of Comprehensive Integrative Medicine, Co-chair of Medical Advisory Team of Healing ALS
Locations (1):
- Virtual, Park City, Utah, United States

IPD SHARING:
Plan to Share IPD: Yes
Individual participant data that underlie the results reported in the published article, after de-identification (text, tables, figures and appendices)
Supporting Information: Study Protocol, CSR
Time Frame: The investigators will share IPD starting 1 year after publication and will make it available for 3 years from that date.
Access Criteria: Researchers who provide a methodologically sound proposal as assessed by our Scientific Advisory Team.
URL: https://HealingALS.org.

REFERENCES:
- [Background] Shochey C. Perimenopause and heavy menstrual flow: standard treatments and alternative treatment modalities. Nurse Pract. 1994 Sep;19(9):73-5. No abstract available. PMID 7816375
- [Background] Brown GC. Rate control within the Na+/glucose cotransporter. Biophys Chem. 1995 Apr;54(2):181-9. doi: 10.1016/0301-4622(94)00132-4. PMID 7756568
- [Background] Ruppert PH, Clemens LG. The role of aromatization in the development of sexual behavior of the female hamster (Mesocricetus auratus). Horm Behav. 1981 Mar;15(1):68-76. doi: 10.1016/0018-506x(81)90035-0. No abstract available. PMID 7216189
- [Background] Arntzen CJ, Dilley RA, Peters GA, Shaw ER. Photochemical activity and structural studies of photosystems derived from chloroplast grana and stroma lamellae. Biochim Biophys Acta. 1972 Jan 21;256(1):85-107. doi: 10.1016/0005-2728(72)90165-x. No abstract available. PMID 4400386
- [Background] Fiore M, Parisio R, Filippini T, Mantione V, Platania A, Odone A, Signorelli C, Pietrini V, Mandrioli J, Teggi S, Costanzini S, Antonio C, Zuccarello P, Oliveri Conti G, Nicoletti A, Zappia M, Vinceti M, Ferrante M. Living near waterbodies as a proxy of cyanobacteria exposure and risk of amyotrophic lateral sclerosis: a population based case-control study. Environ Res. 2020 Jul;186:109530. doi: 10.1016/j.envres.2020.109530. Epub 2020 Apr 15. PMID 32335431
- [Background] Sales de Campos P, Olsen WL, Wymer JP, Smith BK. Respiratory therapies for Amyotrophic Lateral Sclerosis: A state of the art review. Chron Respir Dis. 2023 Jan-Dec;20:14799731231175915. doi: 10.1177/14799731231175915. PMID 37219417
- [Background] Li JY, Sun XH, Cai ZY, Shen DC, Yang XZ, Liu MS, Cui LY. Correlation of weight and body composition with disease progression rate in patients with amyotrophic lateral sclerosis. Sci Rep. 2022 Aug 2;12(1):13292. doi: 10.1038/s41598-022-16229-9. PMID 35918363
- [Background] Bond L, Ganguly P, Khamankar N, Mallet N, Bowen G, Green B, Mitchell CS. A Comprehensive Examination of Percutaneous Endoscopic Gastrostomy and Its Association with Amyotrophic Lateral Sclerosis Patient Outcomes. Brain Sci. 2019 Sep 4;9(9):223. doi: 10.3390/brainsci9090223. PMID 31487846
- [Background] Floeter MK, Mills R. Progression in primary lateral sclerosis: a prospective analysis. Amyotroph Lateral Scler. 2009 Oct-Dec;10(5-6):339-46. doi: 10.3109/17482960903171136. PMID 19922121
- [Background] Syrow L, Calderwood D, Newton C; An Integrative Medicine approach may slow disease in ALS patients compared to standard of care: A pilot observational study. Annals of Neurology Volume 96, Number S32, 149th Annual Meeting American Neurological Association pp. S278-279 (September 2024) https://onlinelibrary.wiley.com/doi/10.1002/ana.27051
- [Background] Harrison D, Mehta P, van Es MA, Stommel E, Drory VE, Nefussy B, van den Berg LH, Crayle J, Bedlack R; Pooled Resource Open-Access ALS Clinical Trials Consortium. "ALS reversals": demographics, disease characteristics, treatments, and co-morbidities. Amyotroph Lateral Scler Frontotemporal Degener. 2018 Nov;19(7-8):495-499. doi: 10.1080/21678421.2018.1457059. Epub 2018 Apr 2. PMID 29607695
- [Background] Crayle J, Lutz M, Raymond J, Mehta P, Bedlack R. Study of "ALS reversals": LifeTime environmental exposures (StARLiTE). Amyotroph Lateral Scler Frontotemporal Degener. 2023 Feb;24(1-2):54-62. doi: 10.1080/21678421.2022.2090846. Epub 2022 Jul 1. PMID 35775279